CLINICAL TRIAL: NCT00795574
Title: Phase 2 Study to Assess the Safety and Efficacy of Infliximab for the Treatment of Hidradenitis Suppurativa
Brief Title: Study to Assess the Safety and Efficacy of Infliximab to Treat Hidradenitis Suppurtativa
Acronym: HS2006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida Academic Dermatology Centers (Other)
Responsible Party: Francisco A Kerdel,M.D., Florida Academic Dermatology Centers
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS2006
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- infliximab (Experimental): Double blind placebo cross-over
  Interventions: Drug: infliximab; Drug: Placebo Comparator
- Placebo (Placebo Comparator): Double blind placebo controlled cross-over
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: infliximab — Dosing is 5mgs/kg at weeks 0,2 and 6 to complete loading dose of drug and then every 8 weeks thereafter until end of treatment phase.
  Arms: infliximab
Drug: Placebo Comparator — 5mgs /kg given IV over a minimum of 2 hours at weeks 0,2 and 6 to complete loading dose and then every 8 weeks during maintenance treatment period.

SUMMARY:
A study to assess the safety and efficacy of the IV drug infliximab for the treatment of hidradenitis suppurativa

ELIGIBILITY:
Inclusion Criteria:

* Person must have moderate to severe Hidradenitis suppurativa
* Multiple ER or doctors visits related to HS
* Intralesional kenalog injection >5/year, but none within 3 months of entry
* HS >1 year duration
* Failed systemic retinoids, but not within 3 months of entry
* Failed at least one prior course of antibiotic therapy, which must not have been administered within 3 months of entry to the study (excluding the recommended antibiotic regimen given immediately before randomization for evidence of active infection
* History of surgery (reconstructive), but not within 3 months of entry

Exclusion Criteria:

* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion (this includes father's who plan on fathering a child within 6 months after their last infusion
* Known allergy against infliximab
* Use of other systemic anti-inflammatory medication except NSAIDs and low dose systemic steroids (equal or less than 10 mg daily prednisolone or equivalent).
* Have had any previous treatment with monoclonal antibodies or antibody fragments.
* Have a known history of serious infections (eg, hepatitis, pneumonia or pyelonephritis) in the previous 3 months.
* Have or have had an opportunistic infection (eg, herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Are considered ineligible according to the TB eligibility assessment, screening, and early detection of reactivation rules defined in Section 26 on: Tuberculosis Eligibility Assessment, Screening, and Early Detection of Reactivation Rules.
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly.
* Currently have any known malignancy or have a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Kerdel, M.D, Principal Investigator — Florida Acadecmic Dermatology Center
Locations (1):
- Florida Academic Dermatology Center, Miami, Florida, United States

REFERENCES:
- [Derived] Grant A, Gonzalez T, Montgomery MO, Cardenas V, Kerdel FA. Infliximab therapy for patients with moderate to severe hidradenitis suppurativa: a randomized, double-blind, placebo-controlled crossover trial. J Am Acad Dermatol. 2010 Feb;62(2):205-17. doi: 10.1016/j.jaad.2009.06.050. PMID 20115947